CLINICAL TRIAL: NCT00922870
Title: Evaluation of Hemodynamic Effects of Cascade Hemofiltration in Septic Shock
Acronym: Cascade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Gambro Lundia AB (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1450
Record Dates: First submitted 2009-06-15; First posted 2009-06-17 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Lasers, Semiconductor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard treatment (Active Comparator)
  Interventions: Other: Standard treatment
- Cascade (Experimental)
  Interventions: Device: Cascade

INTERVENTIONS:
Device: Cascade — Cascade treatment over 48h
  Arms: Cascade
Other: Standard treatment — Standard therapy
  Arms: Standard treatment

SUMMARY:
Septic shock is a major cause of mortality and morbidity in critically ill patients. Septic Shock is associated with an overwhelming, systemic overflow of pro inflammatory and anti-inflammatory mediators, which leads to generalized endothelial damage, multiple organ failure, and altered cellular immunological responsiveness. Although our understanding of the complex pathophysiological alterations that occur in septic shock has increased greatly as a result of recent clinical and preclinical studies, mortality associated with the disorder remains unacceptably high, ranging from 30% to 50%. To date, attempts to improve survival with innovative, predominantly anti-inflammatory therapeutic strategies have been disappointing. A standard hemofiltration rate of 35 ml/kg/hour has been successfully used to treat acute renal failure. However, this dose does not alter plasma levels of inflammatory mediators, suggesting that its ability to clear these mediators is suboptimal. Higher doses of hemofiltration (up to 120 ml/kg per hour) have been demonstrated to improve cardiac function and hemodynamics in several animal models of sepsis. High-volume hemofiltration (HVHF) was thus conceived and applied in patients with septic shock, showing an improvements in hemodynamics with decreased vasopressor requirements and improved survival in patients admitted after a cardiac arrest.

The main benefit described with high volume hemofiltration is a hemodynamic improvement (e.g reduction in catecholamines' requirement). This improvement seems to be due to the removal of a badly defined network of middle molecular weight peptides. To remove efficiently these middle molecular peptides, a high filtration rate is needed. However, with high filtration rates, there is also a high clearance for smaller molecules, including antibiotics, electrolytes, vitamins, trace elements and amino acids.

The cascade hemofiltration system has been designed for a more efficient removal of middle molecular weight peptides with a limited solute consumption.

The goal of this study is the evaluation of the hemodynamic improvement using cascade hemofiltration in patients treated for septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a septic shock diagnosed by the medical staff team.
* Patient mechanically ventilated and treated by high doses of catecholamines after adequate fluid administration (≥ 1.0 mg/h of norepinephrine or epinephrine) for ≥ 120 minutes and < 24h.

Exclusion Criteria:

* Age (years) < 18 or > 85.
* Weight >120 kg
* Thrombocytopenia 50< G/l or Neutrophils <0.5 Giga/l
* Contra indication to heparin anticoagulation.
* Patient requiring catecholamines (epinephrine ≥ 1 mg/h or norepinephrine ≥ 1 mg/h) for >24h.
* Patient admitted to the ICU ≥ 7 days before the inclusion criteria.
* Comorbid conditions with an expected survival < 6 months
* Inclusion (<28 days) in another study interfering with the goals of the current investigation.
* Pregnancy
* Immune compromised patients (e.g. being treated for cancer, treated by immunosuppressors or steroids, AIDS).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
the primary outcome will be the number of days without catecholamines at the 28th day of randomization | 28th day

SECONDARY OUTCOMES:
rate of decrease of catecholamines during the first 72h, days without mechanical ventilation at D90, days without RRT for acute renal failure at D90, days without ICU requirement at D90, status at D90. | 72h, D90

CONTACTS AND LOCATIONS:
Overall Officials: Monchi Mehran, Dr, Study Chair — Unaffiliate
Locations (5):
- France (5):
  - CHU hospital, Clermont-Ferrand
  - Hopital Le Bocage, Dijon
  - Centre Hospitalier Marc JACQUET, Melun
  - Hopital Tenon, Paris
  - Hopital Delafontaine, Saint-Denis